CLINICAL TRIAL: NCT03349892
Title: Stereotactic Ablative Radiotherapy (SABR) for Refractory Ventricular Tachycardia - a Phase I/II Study
Brief Title: Stereotactic Ablative Radiotherapy for Refractory Ventricular Tachycardia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Robert K. Chin, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cardiac SABR
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Results first posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-10

CONDITIONS: Refractory Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Stereotactic Ablation Treatment Arm (Experimental): This is a single-arm, non-blinded study.
  Interventions: Radiation: Stereotactic Ablative Radiotherapy (SABR)

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy (SABR) — A single fraction of radiation is delivered using a clinical radiotherapy system capable of stereotactic radiotherapy to the chest, with on-board image guided radiotherapy capabilities, respiratory motion management, and Intensity Modulated Radiotherapy Treatment (IMRT) planning.
  Other Names: external beam radiation

SUMMARY:
Single arm, phase Ib/2a dose escalation study with an expansion cohort to determine the maximal tolerated dose (MTD) for stereotactic ablative radiotherapy of targets in the cardiac myocardium and to make a preliminary assessment of the efficacy of the treatment. The dose escalation will be guided by Time-to-Event Continual Reassessment Method (TITE-CRM) to ensure more patients will be spared dose limiting toxicities and more patients will be entered on the dose level that will be chosen as minimal dose of maximal effect. This design also allows for continual accrual of patients when delayed adverse events may be observed.

ELIGIBILITY:
Inclusion Criteria:

Documented sustained ventricular arrhythmias refractory to or not a suitable candidate for catheter based RFA ablative therapy

* Documented sustained ventricular arrhythmias refractory to or not a suitable candidate for cardiac sympathetic denervation therapy
* Documented ventricular arrhythmias refractory to or not a suitable candidate for cardiac transplantation
* Documented sustained ventricular arrhythmias refractory to or not a suitable candidate for additional medical management
* ICD in place with documented episodes recurrent VT despite best clinical management previous refusal of ICD with recurrent sustained ventricular arrhythmias
* If ischemic cardiomyopathy, myocardial infarction occurred more than one month prior to enrollment
* No history of prior radiotherapy to the chest
* Prescribed dose must be deliverable using SABR technique
* Age ≥ 18 years
* Karnofsky Performance Status (KPS) > 70
* If a woman is of childbearing potential, a negative serum pregnancy test must be documented. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) for at least 4 weeks after study treatment.
* Ability to understand and willingness to sign a written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Department of Radiation Oncology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stereotactic Ablation Treatment Arm
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Documented sustained ventricular arrhythmias refractory to or not suitable for cardiac transplantation, cardiac sympathetic denervation therapy, catheter based RFA ablative therapy or other medical management.
Arm/Group | Stereotactic Ablation Treatment Arm
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: ICD (Implantable Cardioverter Defibrillator) Shock Free Survival
Description: ICD (implantable cardioverter defibrillator) shock free survival at six months
Time Frame: 6 months
Population: Patients with refractory VT.
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Ablation Treatment Arm
Number analyzed (Participants) | 1
Participants | 1

2. Primary Outcome: Incidence of Salvage Definitive Anti-arrhythmia Therapy (Cardiac Transplant)
Description: Incidence of salvage definitive anti-arrhythmia therapy (cardiac transplant) over 5 years.
Time Frame: 5 years
Population: Single participant was lost to followup prior to 5-year assessment
Arm/Group | Stereotactic Ablation Treatment Arm
Number analyzed (Participants) | 0

3. Secondary Outcome: Incidence of Return of Ventricular Tachycardia Requiring Defibrillation, Intravenous Drug Therapy or Readmission to Hospital
Description: Incidence of return of ventricular tachycardia requiring defibrillation, intravenous drug therapy or readmission to hospital over 5 years
Time Frame: 5 years
Population: Study participant was lost to follow-up prior to 5-year assessment
Arm/Group | Stereotactic Ablation Treatment Arm
Number analyzed (Participants) | 0

4. Secondary Outcome: Incidence of ICD Shocks
Description: Incidence of ICD shocks 12 months post-SABR procedure
Time Frame: 12 months post-SABR procedure
Population: Subject was followed for 28 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Ablation Treatment Arm
Number analyzed (Participants) | 1
Participants | 1

5. Other Pre Specified Outcome: Incidence of Decline of LV Ejection Fraction by More Than 5% on Two Consecutive Echocardiograms
Description: Incidence of decline of LV ejection fraction by more than 5% on two consecutive echocardiograms over 5 years
Time Frame: 5 years
Population: Subject was not followed for 5 years
Arm/Group | Stereotactic Ablation Treatment Arm
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Incidence of Persistent Increase in Baseline Supplemental Oxygen Requirement by 1L for a Duration of >3 Months
Description: Incidence of persistent increase in baseline supplemental oxygen requirement by 1L for a duration of >3 months over 5 years
Time Frame: 5 years
Population: Subject was not followed for 5 years
Arm/Group | Stereotactic Ablation Treatment Arm
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Incidence of Steroid Use for Radiotherapy Related Indications
Time Frame: 5 years
Population: Subject was not followed for 5 years
Arm/Group | Stereotactic Ablation Treatment Arm
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Overall Survival
Time Frame: Followed for 10 years +
Population: Subject was not followed for 10 years
Arm/Group | Stereotactic Ablation Treatment Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 28 months
Arm/Group | Stereotactic Ablation Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT03349892/Prot_SAP_000.pdf